CLINICAL TRIAL: NCT05026229
Title: A Randomized Controlled Study of Dasatinib Combined With Reduced Intensive Consolidation Chemotherapy in Newly Diagosed Philadelphia Chromesome Positive Adult Lymphoblastic Leukemia
Brief Title: A Study of Dasatinib Plus Reduced Intensive Consolidation Chemotherapy in Ph+ Adult ALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2020-002-2
Record Dates: First submitted 2021-08-17; First posted 2021-08-30 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-08

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia-Positive Acute Lymphoblastic Leukemia; ALL, Adult
Keywords: Philadelphia-Positive; Adult Acute Lymphoblastic Leukemia; Tyrosine Kinase Inhibitor; Consolidation Chemotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib; Consolidation Chemotherapy; Vincristine; Prednisone; VDA-P protocol; Methotrexate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dasatinib, Vincristine and Prednisone (Experimental): After induction therapy, the patients in the 'Dasatinib, Vincristine and Prednisone' group will receive dasatinib and consolidation chemotherapy with vincristine and prednisone.
  Interventions: Drug: dasatinib plus consolidation chemotherapy with vincristine and prednisone
- Dasatinib, Methotrexate and Cytarabine (Experimental): After induction therapy, the patients in the 'Dasatinib, Methotrexate and Cytarabine' group will receive dasatinib and consolidation chemotherapy with high-dose methotrexate and cytarabine.
  Interventions: Drug: dasatinib plus consolidation chemotherapy with high-dose methotrexate and cytarabine

INTERVENTIONS:
Drug: dasatinib plus consolidation chemotherapy with vincristine and prednisone — After induction therapy, the patients in the 'Dasatinib, Vincristine and Prednisone' group will receive dasatinib and consolidation chemotherapy with vincristine and prednisone.
  Other Names: Dasatinib + VP Regimen
  Arms: Dasatinib, Vincristine and Prednisone
Drug: dasatinib plus consolidation chemotherapy with high-dose methotrexate and cytarabine — After induction therapy, the patients in the 'Dasatinib, Methotrexate and Cytarabine' group will receive dasatinib and consolidation chemotherapy with high-dose methotrexate and cytarabine.
  Other Names: Dasatinib + HyperB Regimen
  Arms: Dasatinib, Methotrexate and Cytarabine

SUMMARY:
This project is a key clinical research project approved by the Clinical Research Center of the First Affiliated Hospital of Xi'an Jiaotong University. Tyrosine kinase inhibitors (TKI) combined with intensive chemotherapy has markedly improved the outcomes of philadelpha-positive lymphoblastic leukemia (Ph+ ALL). However, a considerable proportion of patients failed to complete the intended chemotherapy and some even died early. The optimal balance between the intensity of chemotherapy and safety should be explored. In this study, Ph+ ALL patients who achieve complete remission (CR) after VP regimen (vincristine and prednisone) plus dasatinib as induction are enrolled and then the participants will receive different consolidation chemotherapy. Patients in the group A will continue to use VP regimen plus dasatinib, while the group B receives hyper-CVAD/methotrexate-cytarabine regimen plus dasatinib. The measurable residual disease (MRD), CR, adverse effects (AE), overall survival (OS) and disease free survival (DFS) will be observed to determine the proper consolidation chemotherapy regimen.

DETAILED DESCRIPTION:
About 25% of adult patients with acute lymphoblastic leukemia (ALL) are associated with t (9; 22), positive philadelphia chromosome (Ph+ ALL), in whom BCR/ABL fusion gene can be detected in the bone marrow and peripheral blood. The use of tyrosine kinase inhibitors (TKI) plus intensive chemotherapy has markedly improved the outcomes of Ph+ ALL. However, it's reported that 74% pf patients failed to complete the intended chemotherapy, and early death occured in a considerable proportion of patients during induction. The optimal balance between the intensity of chemotherapy and safety need to be explored. In this study, Ph+ ALL patients are enrolled. The participants will receive dasatinib and induction chemotherapy using VP regimen (vincristine and prednisone) to achieve complete remission (CR). Then the participants will be randomly divided into two groups. The subjects inthe group A will continue to use VP regimen plus dasatinib as consolidation, while the patients in the group B receive hyper-CVAD/methotrexate-cytarabine regimen plus dasatinib. The measurable residual disease (MRD), CR, adverse effects (AE), overall survival (OS) and disease free survival (DFS) will be observed to determine the proper consolidation chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old, newly diagnosed as Ph+ALL.
* Sign the informed consent.
* Accept consolidation chemotherapy.
* Accept follow-up.

Exclusion Criteria:

* Liver and kidney function impairment: serum transaminase > 2 times of the upper limit of normal value, total bilirubin > 1.5 times of the upper limit of normal value, serum inosine > the upper limit of normal value (97 umol/L).
* Active hepatitis B, hepatitis C or tuberculosis infection.
* Can not tolerate the adverse effects of dasatinib.
* Pregnancy.
* Diagnosis of mental disorders.
* Do not accept follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Measurable Residual Disease (MRD) Positivity | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  MRD refers to the subclinical levels of residual leukemia.
Percentage of Participants with Complete Remission (CR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  CR means that the blood counts have returned to normal, the leukemia cannot be seen when a bone marrow sample is examined under the microscope, and the signs and symptoms of the ALL are gone.

SECONDARY OUTCOMES:
disease-free survival (DFS), months | From date of consolidation chemotherapy until disease progression, the end of follow-up or the date of death from any cause, whichever came first.
  The measure of time after consolidation chemotherapy during which no sign of ALL is found.
overall survival (OS), months | From date of consolidation chemotherapy until the end of follow-up or the date of death from any cause, whichever came first.
  The length of time from the date of diagnosis that Ph+ ALL patients are still alive.
adverse effects (AE) | From date of consolidation chemotherapy until the end of follow-up or the date of death from any cause, whichever came first.
  An adverse effect is any untoward medical occurrence in clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pengcheng He, Study Chair — First Affiliated Hospital of Xian Jiaotong University; Xiaoning Wang, Study Director — First Affiliated Hospital of Xian Jiaotong University; Huachao Zhu, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University; Juan Ren, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University; Ying Chen, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University; Ting Fan, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China